CLINICAL TRIAL: NCT02701868
Title: Unintentional Overfeeding of Formula Fed Infants
Acronym: Whoa Baby
Status: Completed | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Anne Gilmore, Postdoctoral Fellow, Pennington Biomedical Research Center
Other Study IDs: PBRC2016-002
Record Dates: First submitted 2016-02-22; First posted 2016-03-08 (Estimated); Results first posted 2021-01-14 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2020-12

CONDITIONS: Childhood Obesity; Infant Development
Keywords: Infant Formula
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Phase 1: Up to 40 individuals will be recruited to participate in focus groups at Pennington Biomedical Research Center. Approximately six focus groups (each with 5-10 participants) will be conducted at the Pennington Biomedical Demonstration Kitchen over the course of approximately 3 months.
- Phase 2: Up to 150 individuals who did not participate in Whoa Baby Phase 1 will be recruited to test the efficacy of the revised instructions on infant overfeeding in comparison with the instructions currently provided on the packaging.

SUMMARY:
Although breast milk is recommended exclusively until 6 months of age, two-thirds of infants in the U.S. are fed infant formula. Despite an almost identical energy density between infant formula and breast milk, formula fed infants experience greater weight gain in the first year of life. The investigators propose that unintentional overfeeding, of nearly one additional day of calories per week, due to the "over-scooping" of powdered formula contributes significantly to this phenomenon and potentially to the early development of childhood obesity, a significant public health problem.

DETAILED DESCRIPTION:
In the proposed study the investigators will assess the literacy and understanding of individuals to follow commercially available infant formula instructions. The investigators will collaborate with the LA CaTS Health Literacy Core to improve the reading and comprehension of the manufacturer package instruction, and will solicit the input of caregivers and key stakeholders to inform the development of educational intervention around infant feeding. Following modification of infant formula preparation instructions, the investigators will conduct a randomized controlled trial that will test the efficacy of the modified instructions on infant overfeeding in comparison with the manufacturer package instructions. One hundred and fifty participants will be asked to complete one study visit during which they will be asked to measure various serving sizes of infant formula following either the manufacturer package instructions or the modified instructions.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Willing to participate in 1 assessment visit at Pennington Biomedical Research Center
* English speaking

Exclusion Criteria:

* <18 years of age
* Not willing to participate in 1 assessment visit at Pennington Biomedical Research Center
* Non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Up to 40 individuals will be recruited to participate in focus groups at Pennington Biomedical Research Center. Phase 1 will utilize qualitative data gathered from focus groups to direct the modification of infant formula manufacturer preparation instructions to enhance user understanding and accuracy. The modified instructions will be used in Phase 2.
  Up to 150 individuals will be enrolled in Phase 2 to test the efficacy of the revised instructions on infant overfeeding in comparison with the instructions currently provided on the packaging.
Sampling Method: Probability Sample
Enrollment: 171 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Gilmore, Ph.D., Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1: Up to 40 individuals will be recruited to participate in focus groups at Pennington Biomedical Research Center. Approximately six focus groups (each with 5-10 participants) will be conducted at the Pennington Biomedical Research Center Demonstration Kitchen over the course of approximately 3 months.
- Phase 2 Standard Instructions: Up to 150 individuals who did not participate in Whoa Baby Phase 1 will be recruited for Phase 2. Up to 75 individuals will be randomized to prepare infant formula using standard instructions.
- Phase 2 Modified Instructions: Up to 150 individuals who did not participate in Whoa Baby Phase 1 will be recruited for Phase 2. Up to 75 individuals will be randomized to prepare infant formula using modified instructions.
Period: Overall Study
Arm/Group | Phase 1 | Phase 2 Standard Instructions | Phase 2 Modified Instructions
Started | 21 | 75 | 75
Completed | 21 | 75 | 75
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase 2 Standard Instructions: Up to 75 individuals who did not participate in Whoa Baby Phase 1 were recruited to prepare bottles using the standard infant formula preparation instructions.
- Phase 2 Modified Instructions: Up to 75 individuals who did not participate in Whoa Baby Phase 1 were recruited to prepare bottles using the modified infant formula preparation instructions. The modified instructions were developed as a result of the focus groups' conditions in Phase 1.
- Total: Total of all reporting groups
Arm/Group | Phase 1 | Phase 2 Standard Instructions | Phase 2 Modified Instructions | Total
Number analyzed (Participants) | 21 | 75 | 75 | 171
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.5 (11.7) | 36.0 (15.8) | 40.6 (17.6) | 37.8 (16.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 65 | 59 | 141
  Male | 4 | 10 | 16 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 0 | 3 | 4 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 6 | 25 | 15 | 46
  White | 15 | 46 | 54 | 115
  More than one race | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 1 | 1
BMI, Continuous [Mean (Standard Deviation); unit: kg/m^2] | 26.8 (8.1) | 29.6 (6.6) | 29.5 (7.9) | 29.2 (7.5)
Education, Categorical [Count of Participants; unit: Participants]
  High School Diploma/GED or Less | 1 | 8 | 5 | 14
  1-3 Years College | 5 | 26 | 37 | 68
  College Degree | 9 | 25 | 17 | 51
  Post-Graduate Degree | 6 | 16 | 16 | 38
Income, Categorical [Count of Participants; unit: Participants]
  <$30,000/year | 5 | 21 | 21 | 47
  $30,000-$99,999/year | 9 | 32 | 28 | 69
  >$80,000/year | 7 | 21 | 25 | 53
  No answer | 0 | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Focus Group Recommendations to Improve Infant Formula Preparation Instructions
Description: Focus groups were used to evaluate and provide recommendations to improve the reading and comprehension of powdered infant formula package preparation instructions. Five focus groups provided primary recommendations. The percentage of focus group participants reporting specific recommendations are summarized.
Time Frame: Day 1
Population: The focus groups were only completed for Phase 1 participants. This outcome measure does not apply to Phase 2 participants who did not participate in focus groups and provide infant formula preparation instructions.
Measure: Number; unit: percentage of focus group participants
Arm/Group | Phase 1 | Phase 2
Number analyzed (Participants) | 21 | 0
percentage of focus group participants
  Pictures were helpful | 60 |
  Clarify Safety Information | 80 |
  Define and emphasize "level" and "unpacked" scoop | 100 |
  Move mixing guide to the top | 60 |

2. Primary Outcome: Percent Error of Dispensed Formula Weight as Compared to Expected Formula Weight
Description: Percent Error of the formula weight prepared by Phase 2 study participants as compared to the expected formula weight from the manufacturer's label. Phase 2 participants were either randomly assigned the standard instructions or the instructions that were modified as a result of the Phase 1 focus groups.
  Percent error was calculated as the measured formula weight prepared by Phase 2 study participants subtracted from the expected formula weight found on the manufacturer's label with that result being divided by the expected formula weight found on the manufacturer's label. The final result is multiplied by 100 to provide the percent error. Percent error is presented as opposed to formula weight because each participant prepared two 2, 4, 6, and 8 oz bottles. Percent error analysis includes all bottles prepared regardless of size.
Time Frame: Day 1
Population: This outcome measure does not apply to Phase 1 participants because Phase 1 participants did not participate in the double blind, randomized controlled portion of the trial. Phase 1 participants did not prepare infant formula bottles according to either the standard or modified instructions.
Measure: Mean (Standard Deviation); unit: percentage of error
Arm/Group | Phase 1 | Phase 2 Standard Instructions | Phase 2 Modified Instructions
Number analyzed (Participants) | 0 | 75 | 75
percentage of error |  | -4.66 (0.74) | -0.67 (0.76)

ADVERSE EVENTS:
Time Frame: 1 day
Description: Adverse event data were not collected systematically as part of study data, but reported by study participants as applicable.
Arm/Group | Phase 1 | Phase 2 Standard Instructions | Phase 2 Modified Instructions
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/75 | 0/75
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/75 | 0/75
Other Adverse Events (participants affected / at risk) | 0/21 | 0/75 | 0/75

LIMITATIONS AND CAVEATS:
This study involved two phases: Phase 1 was participatory research where participants were involved in focus groups and Phase 2 was a double-blind randomized controlled trial where participants were randomly assigned to prepare infant formula bottles using the standard manufacturer's instructions or the instructions that were modified as a result of Phase 1 focus groups. Due to the design, primary outcomes were different for Phase 1 and Phase 2. Both primary outcomes are included in the results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-28): https://cdn.clinicaltrials.gov/large-docs/68/NCT02701868/Prot_SAP_000.pdf